CLINICAL TRIAL: NCT00549458
Title: Randomized Controlled Trial Comparing Traditional Pelvic Floor Rehabilitation to Pilates in Increasing Pelvic Muscles Strength.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Patrick Culligan, MD, Atlantic Urogynocology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AH Urogynecology
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Muscle Weakness
Keywords: Week pelvic floor muscle in females
MeSH Terms: conditions — Muscle Weakness | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Pilates — The currently popular exercise program, known as Pilates (named after founder, Joseph Pilates) consists of a series of low impact, flexibility and muscle toning exercises. The philosophy centers around developing core strength which includes strengthening the pelvic floor. Its use has been described in the US since the 1920s.4 Five million Americans currently participate, as opposed to five thousand ten years ago.5 Given its mainstream popularity, Pilates would be an appealing as a therapeutic modality for women experiencing pelvic muscle weakness. Currently, there are no studies that assess the efficacy of Pilates in increasing pelvic muscle strength.
Procedure: Pelvic muscle rehabilitation therapy — The currently popular exercise program, known as Pilates (named after founder, Joseph Pilates) consists of a series of low impact, flexibility and muscle toning exercises. The philosophy centers around developing core strength which includes strengthening the pelvic floor. Its use has been described in the US since the 1920s.4 Five million Americans currently participate, as opposed to five thousand ten years ago.5 Given its mainstream popularity, Pilates would be an appealing as a therapeutic modality for women experiencing pelvic muscle weakness. Currently, there are no studies that assess the efficacy of Pilates in increasing pelvic muscle strength.

SUMMARY:
The objective of this randomized controlled trial is to determine whether a standardized Pilates exercise program can effectively strengthen pelvic floor muscles when compared with conventional pelvic muscle rehabilitation.

Urinary incontinence is a widespread problem that affects 10-40% of all ambulatory women and pelvic floor muscle training is an effective treatment for this problem. However, its efficacy is proportionate to the effort expended. Even among women who are diligent with pelvic muscle rehabilitation, long term follow-up reveals that benefits are lost in the absence of maintenance exercises.

While this intervention is effective, recent studies demonstrate that long term adherence to treatment is low. As compliance appears to be a prerequisite to achieving sustained benefit, finding a method of pelvic muscle strengthening that better lends itself to long term commitment could prove beneficial.

The currently popular exercise program, known as Pilates (named after founder, Joseph Pilates) consists of a series of low impact, flexibility and muscle toning exercises. The philosophy centers around developing core strength which includes strengthening the pelvic floor. Its use has been described in the US since the 1920s.4 Five million Americans currently participate, as opposed to five thousand ten years ago.5 Given its mainstream popularity, Pilates would be an appealing as a therapeutic modality for women experiencing pelvic muscle weakness. Currently, there are no studies that assess the efficacy of Pilates in increasing pelvic muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 yrs or older

Exclusion Criteria:

* Pregnancy
* No pelvic organ prolapse beyond the hymenal ring.
* Age or medical condition that make it difficult for patient to tolerate exam or follow verbal instructions.
* Pacemakers
* IUDs
* Vaginal infections or urinary tract infections
* Medical or physical conditions which exclude the proper performance of Pilates.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Increase pelvic floor strength | Over a 12 week period of time

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Culligan, MD, Principal Investigator — Atlantic Health Urogynecology
Locations (1):
- Office of Urogynecolgy 95 Madison Avenue Suite 204, Morristown, New Jersey, United States